CLINICAL TRIAL: NCT05154513
Title: Long-Term Clinical, Immunologic, and Virologic Profiles of Children Who Received Early Treatment for HIV
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT 2028; 5UM1AI068632-19 (NIH); HHSN275201800001I (Other Grant/Funding Number: Eunice Kennedy Shriver National Institute of Child Health and Human Development)
Record Dates: First submitted 2021-03-04; First posted 2021-12-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following specimens will be collected: HIV-1 RNA PCR, HIV-1 DNA ddPCR, CD4+ and CD8+ cell counts and percentages, HIV-1 antibody, Serum, plasma, and peripheral blood mononuclear cell (PBMC) storage, ARV resistance testing if clinically indicated. If child is three years of age or older, collect nasopharyngeal and rectal swabs for storage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Children living with perinatally-acquired HIV who received early treatment in IMPAACT network studies or other research studies sponsored by the United States National Institutes of Health.
  Interventions: Other: Cohort 1

INTERVENTIONS:
Other: Cohort 1 — No intervention provided in this study

SUMMARY:
IMPAACT 2028 is an observational prospective study to characterize a cohort of early treated children who may participate in future research related to HIV remission or cure. Up to approximately 250 participants will be in the study for approximately seven years. No intervention is provided in the study.

DETAILED DESCRIPTION:
This is an observational prospective cohort study characterizing and establishing a biorepository of early treated children who may participate in future research related to HIV remission or cure. Early treatment is defined as treatment with at least three ARV agents from at least two classes of ART initiated within 12 weeks of birth. Within the overall study population, for descriptive and analysis purposes, children who initiated treatment within 48 hours of birth will be classified as having received very early treatment. A subset of children will have received bNAbs as part of their treatment regimens.

Up to approximately 250 children living with HIV who received early treatment in IMPAACT network studies or other research studies sponsored by the US National Institutes of Health (NIH) will be enrolled and followed semi-annually for up to seven years. Clinical, virologic, and immunologic evaluations will be performed semi-annually at each study visit, and specimens will be collected for the study's biorepository for future investigations.

ELIGIBILITY:
Inclusion Criteria:

* Participated in one of the parent studies
* Confirmed HIV-1 infection based on documented nucleic acid testing of two blood samples collected at different time points
* Received early treatment for HIV-1 infection, defined as treatment with at least three ARV agents from at least two classes of ART, initiated within 12 weeks of birth
* Based on parent or guardian report at entry, child is expected to be available for at least 24 months of follow-up
* Parent or guardian is willing and able to provide written informed consent for child's study participation and, when applicable per institutional review board/ethics committee (IRB/EC) policies and procedures, child is willing and able to provide written assent for study participation

Exclusion Criteria:

* Has any documented or suspected clinically significant medical condition or any other condition that, in the opinion of the site investigator, would make participation in the study unsafe or otherwise interfere with completing study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to approximately 250 children living with HIV who received early treatment in IMPAACT network studies or other research studies sponsored by the US National Institutes of Health (NIH)
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome Measures - Weight measured in kg | At enrollment, at participant study completion (up until 7 years)
  Median and interquartile range; to characterize long-term clinical profile
Clinical Outcome Measures - Height measured in cm | At enrollment, at participant study completion (up until 7 years)
  Median and interquartile range; to characterize long-term clinical profile
Clinical Outcome Measures - Weight-for-height Z score | At enrollment, at participant study completion (up until 7 years)
  Median and interquartile range, % of participants with Z scores corresponding to mild, moderate, or severe malnutrition
Clinical Outcome Measures - Head circumference measured in cm | At birth, 24 months of age
  Median and interquartile range; to characterize long-term clinical profile
Clinical Outcome Measures - Head circumference-for-age Z score | At birth, 24 months of age
  Median and interquartile range; to characterize long-term clinical profile
Clinical Outcome Measures - Cumulative incidence of WHO clinical Stage 3 or Stage 4 conditions | At enrollment, at participant study completion (up until 7 years)
  % of patients with outcome; to characterize long-term clinical profile
Clinical Outcome Measures - Cumulative incidence of medical conditions that required hospitalization, resulted in persistent or significant disability or incapacity, were life threatening, or resulted in death | At enrollment, at participant study completion (up until 7 years)
  % of patients with outcome; to characterize long-term clinical profile
Clinical Outcome Measures - Cumulative incidence of other medical conditions of interest | At enrollment, at participant study completion (up until 7 years)
  % of patients with outcome; to characterize long-term clinical profile
Clinical Outcome Measures - Cumulative incidence of mortality | At study participant completion (up until 7 years)
  % of patients with outcome; to characterize long-term clinical profile
Immunologic Outcome Measures - CD4+ cell counts and percentages | At enrollment, at participant study completion (up until 7 years)
  Median and interquartile range; to characterize long-term immunologic profile
Immunologic Outcome Measures - CD8+ cell counts and percentages | At enrollment, at participant study completion (up until 7 years)
  Median and interquartile range; to characterize long-term immunologic profile
Immunologic Outcome Measures - HIV-1 antibody status | At enrollment, at participant study completion (up until 7 years)
  % of participants with negative serostatus
Virologic Outcome Measures - HIV-1 RNA in plasma | At enrollment, at participant study completion (up until 7 years)
  % of participants with HIV-1 RNA below the limit of detection of the assay among participants with quantifiable HIV-1 RNA, median and interquartile range
Virologic Outcome Measures - HIV-1 DNA concentration in PBMCs | At enrollment, at participant study completion (up until 7 years)
  % of participants with HIV-1 DNA below the limit of detection of the assay among participants with quantifiable HIV-1 DNA, median and interquartile range
Virologic Outcome Measures - HIV-1 ARV resistance mutations | At enrollment, at participant study completion (up until 7 years)
  % of participants with resistance mutations

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Barnabas, MD, PhD, Study Chair — University of Stellenbosch; Samantha Fry, MD, MMed, Study Chair — University of Stellenbosch; Julia Rosebush, DO, FAAP, Study Chair — University of Chicago
Locations (28):
- United States (6):
  - David Geffen School of Medicine at UCLA (CRS 5112), Los Angeles, California
  - University of Colorado (5052), Aurora, Colorado
  - 5055, South Florida CDTC Fort Lauderdale Clinical Research Site, Fort Lauderdale, Florida
  - Univ of Miami Pediatric/Perinatal HIV/AIDS (5127), Miami, Florida
  - 5030, Emory University School of Medicine Clinical Research Site, Atlanta, Georgia
  - 5128, Texas Children's Hospital Clinical Research Site, Houston, Texas
- Botswana (2):
  - Gaborone CRS 12701, Gaborone
  - Molepolole Prevention/Treatment Trials CRS 12702, Molepolole
- Brazil (5):
  - School of Medicine, University of Minas Gerais - FUNDEP (5073), Belo Horizonte
  - 5071, Instituto de Puericultura e Pediatria Martagao Gesteira Clinical Research Site, Rio de Janeiro
  - Hospital dos Servidores Rio de Janeiro, Rio de Janeiro
  - Hospital Geral De Nova Igaucu (5097), Rio de Janeiro
  - Ribeirao Preto Medical School, University of Sao Paulo (5074), São Paulo
- Les Centres GHESKIO (30022), Port-au-Prince, Haiti
- 5121, Kenya Medical Research Institute/Walter Reed Project Clinical Research Center Kericho Clinical Research Site, Kericho, Kenya
- Malawi (2):
  - College of Med. JHU CRS (30301), Blantyre
  - University of North Carolina Lilongwe (12001), Lilongwe
- South Africa (4):
  - Soweto IMPAACT CRS (8052), Johannesburg, Gauteng
  - 30300, Umlazi Clinical Research Site, Durban
  - 8051, Wits RHI Shandukani Research Centre Clinical Research Site, Johannesburg
  - Family Clinical Research Unit (FAM-CRU) CRS (8950), Tygerberg Hills
- Kilimanjaro Christian Medical Centre (5118), Moshi, Tanzania
- Thailand (2):
  - Siriraj Hospital Mahidol University CRS (5115), Bangkok, Ratchathewi
  - Chiang Rai Regional Hospital (5116), Chiang Rai
- 31798, Baylor-Uganda Clinical Research Site, Kampala, Uganda
- Zimbabwe (3):
  - Seke North CRS 30306, Chitungwiza
  - St. Mary's CRS 30303, Chitungwiza
  - Harare Family Care (31890), Harare

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT05154513/Prot_ICF_000.pdf